CLINICAL TRIAL: NCT07213102
Title: Integration of Household-Based Interventions With Early Childhood Programming: A Randomized Controlled Trial in the Philippines
Brief Title: Transform + Family Academy Randomized Controlled Trial in the Philippines
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Care Ministries, Philippines (Other)
Collaborators: Compassion International, United States of America (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: icmcompassionrct; icmcompassionrct (Other: Compassion)
Record Dates: First submitted 2025-09-25; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Child Development; Child Nutrition, Child Neurobehavioral Development; Household and Family; Financial Wellbeing; Academic Attainment
Keywords: Child Development; Child Nutritional Status; Household Financial Resilience

STUDY DESIGN:
Intervention Model Description: This study is an individual-level randomized controlled trial. A total of 700 households with children aged 3-5 years from Compassion International communities across Western and Southern Mindanao will be randomly assigned to one of two treatment arms: Treatment and Control. The treatment will be assigned at the household level, with community-level and regional-level stratification, to ensure balanced representation across geographic locations.
  Control households will continue receiving Compassion International's Survival and Early Childhood Program. Treatment households will receive an integrated intervention combining Compassion International's Survival and Early Childhood Program with International Care Ministries' Transform + Family Academy program.
  A roster of eligible households will be compiled and randomly allocated to one of two treatment arms. To minimize bias, participant recruitment and enrollment will occur prior to random treatment assignment.
Masking Description: Due to the nature of the interventions, participants cannot be blinded to their treatment assignment as treatment participants will attend Transform + Family Academy sessions while control participants will not. Implementation staff will necessarily know group assignments to deliver appropriate interventions. This is an unblinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment receiving integrated Survival and Early Childhood Program & Transform + Family Academy (Experimental): Treatment: Participants will continue receiving Compassion International's Survival and Early Childhood Program and additionally receive International Care Ministries' Transform + Family Academy program.
  In the treatment arm, the integrated intervention will be delivered over 4 months with participants continuing to receive the Survival and Early Childhood Program. In addition to this, participants receive Transform + Family Academy, with 15 Transform sessions conducted weekly at community locations and 8 weeks of Family Academy sessions delivered through home visits. Each Transform session includes 90-minute health and livelihood training by ICM staff, with optional values components facilitated by community leaders. Family Academy provides home-based early numeracy and phonics lessons for children and their caregivers.
  Interventions: Other: Integrated Whole-Household Programming
- Control receiving standard Survival and Early Childhood Program (Active Comparator): Control: Participants will continue receiving Compassion International's Survival and Early Childhood Program without additional interventions.
  Interventions: Other: Standard Child-Focused Programming

INTERVENTIONS:
Other: Integrated Whole-Household Programming — Treatment participants receive both Compassion International's Survival and Early Childhood Program (holistic child development through health support, educational programming, social development, and spiritual formation via local community partners) plus International Care Ministries' Transform + Family Academy intervention. The Transform component is a 15-week household-level program including health education covering malnutrition prevention, sanitation, respiratory infections, infant care; livelihood training focused on income diversification and business development with savings group formation; and values formation addressing personal character, family relationships, and decision-making. The Family Academy component provides home-based early numeracy and phonics instruction (one hour per topic) to children aged 3-5 with concurrent caregiver capacity building for school readiness support, delivered over 8 weeks.
  Other Names: Whole-household poverty intervention
  Arms: Treatment receiving integrated Survival and Early Childhood Program & Transform + Family Academy
Other: Standard Child-Focused Programming — Compassion International's Survival and Early Childhood Program provides holistic child development through health support, nutritional assistance, educational programming, social development, and spiritual formation delivered via local community partners.
  Arms: Control receiving standard Survival and Early Childhood Program

SUMMARY:
This study evaluates the integration of two complementary poverty alleviation programs: Compassion International's (CI) child-focused Survival and Early Childhood Program with International Care Ministries' (ICM) household-level Transform + Family Academy intervention. CI's program provides holistic child development through health support, educational programming, social development, and spiritual formation via local church partners for children aged 3-5 years. ICM's Transform + Family Academy combines a 15-week household intervention targeting health education, livelihood training, and values formation with an 8-week early childhood education component delivered through home visits.

The primary aim of this research is to assess whether integrating household-level interventions with child-focused programming enhances early numeracy and literacy outcomes among children aged 3-5 living in extreme poverty in Western and Southern Mindanao, Philippines. The study also examines the intervention's impact on children's nutritional status and household financial resilience, including savings behaviors and access to social safety nets.

The investigators hypothesize that addressing household-level constraints including caregiver capacity, health, and economic challenges will enhance children's academic and nutritional outcomes alongside household financial resilience compared to child-focused programming alone.

DETAILED DESCRIPTION:
This individual-level randomized controlled trial examines the integration of Compassion International's (CI) child-focused Survival and Early Childhood Program with International Care Ministries' (ICM) household-level Transform + Family Academy intervention among 700 families with children aged 3-5 years across CI's partner communities in Western and Southern Mindanao, Philippines. All participating households are currently registered in CI's Survival and Early Childhood Program, which provides comprehensive child development support through local community partners. Through random assignment, half of the households will additionally receive ICM's household-level intervention targeting the broader family system.

This study examines whether combining ICM's household-level interventions with CI's child-focused programming can improve developmental outcomes for children aged 3-5 years in extreme poverty settings. The research evaluates the effectiveness of ICM's Transform + Family Academy approach to addressing broader family constraints, including caregiver capacity, health challenges, and economic instability, on children's developmental outcomes and household financial resilience when integrated with CI's Survival and Early Childhood Program. Specifically, the outcomes of interest include children's early numeracy and literacy development, alongside secondary outcomes of children's nutritional status and household financial resilience as measured through savings behaviors and social safety net access.

The hypothesis underlying this work suggests that child development programs may achieve greater impact when paired with comprehensive household support that tackles the multidimensional nature of poverty affecting both immediate child needs and the family systems that sustain long-term progress.

ICM's Transform component is a 15-week program delivered through weekly 90-minute community-based group sessions covering three domains: health education (malnutrition prevention, sanitation, respiratory infections, infant care), livelihood training (income diversification, business development, savings group formation), and values formation (personal character, family relationships, decision-making). Health and livelihood sessions are facilitated by trained ICM staff, while optional values components are delivered by community leaders.

The Family Academy component provides 8 weeks of home-based early childhood education through twice-weekly visits delivering separate one-hour sessions for mathematics and phonics instruction. These sessions target both children aged 3-5 and their caregivers, building caregiver capacity to support school readiness through structured learning activities and educational games.

Eligible households must have a child aged 3-5 currently registered in CI's Survival and Early Childhood Program and meet ICM's poverty criteria (poverty score of 50 or above based on asset-based scoring and household income evaluation). Each household must include an adult caregiver aged 18-65 who can provide informed consent. Households with previous participation in ICM interventions are excluded. Households are individually randomly assigned to treatment groups using stratified randomization by community and regional levels to ensure balanced allocation across geographic locations.

Control households continue receiving CI's standard Survival and Early Childhood Program. Treatment households receive the integrated intervention combining CI's programming with ICM's Transform + Family Academy delivered over four months. All data collection is conducted by trained external enumerators at five timepoints: baseline, pre-Family Academy, post-Family Academy, midline (2 months post-intervention), and endline (12 months post-intervention).

The following analyses will be conducted for the research objectives to assess the impact of the integrated intervention:

Primary:

* Linear regression models with cluster-robust standard errors will analyze differences in children's early numeracy competency composite scores between Treatment and Control groups.
* Linear regression models with cluster-robust standard errors will analyze differences in children's phonics and literacy competency composite scores between Treatment and Control groups.

Secondary:

* Linear regression models with cluster-robust standard errors will analyze differences in children's weight-for-height z-scores between Treatment and Control groups.
* Logistic regression models with cluster-robust standard errors will analyze differences in probability of having household savings between Treatment and Control groups.
* Linear regression models with cluster-robust standard errors will analyze differences in total household savings amounts between Treatment and Control groups.
* Linear regression models with cluster-robust standard errors will analyze differences in social safety net access index scores between Treatment and Control groups.

All models will include baseline outcome measures as covariates and strata fixed effects for randomization stratification (community and regional levels). Analyses will be conducted separately for short-term effects (1 week after intervention and 2-month follow-up) and sustained effects at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Households must have a child between 3 to 5 years old who is currently registered in CI's Survival and Early Childhood Program.
* Households must meet ICM's poverty criteria with a poverty score of 50 and above as determined through asset-based scoring and household income evaluation. Higher scores indicate poorer households.
* Each participating household must include an adult family member aged 18 to 65 years who serves as a primary caregiver for the target child.

Exclusion Criteria:

* Households with previous participation in ICM's Transform program will be excluded from the study.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Children's early numeracy competency at post-intervention and 12 months | Baseline, 1 week after intervention, and 12 months
  Children's early numeracy competency is assessed through proctored assessments testing early learning proficiency using eight subtasks to measure preschool children's early math skills. The assessment measures children's mathematical skills across eight components: color recognition (10 points), shape recognition (8 points), rote count (10 points), object count (10 points), numeral identification (10 points), numeral comparison (9 points), missing number (10 points), and simple addition (10 points). The total possible score is 77 points, with higher scores indicating better numeracy skills.
Children's phonics and literacy competency at post-intervention and 12 months | Baseline, 1 week after intervention, and 12 months
  Children's phonics and literacy competency is assessed through proctored assessments testing pre-reading skills and phonemic awareness. The assessment measures children's reading and phonics skills across four components: alphabet recitation (10 points), letter name identification (20 points), beginning sound recognition (20 points), and letter sound identification (20 points). The total possible score is 70 points, with higher scores indicating better literacy and phonics skills.

SECONDARY OUTCOMES:
Children's malnutrition status at 2 months and 12 months | Baseline, 2 months, and 12 months
  Children's malnutrition status is evaluated through anthropometric measurements where weight-for-height ratios are transformed into standardized z-scores based on World Health Organization reference standards for pediatric populations. Malnutrition in children under 5 years is defined as weight-for-height z-scores below -2 standard deviations in the absence of edema.
Household savings at 2 months and 12 months | Baseline, 2 months, and 12 months
  The household savings measure assesses household financial resources through two indicators: the probability of having savings (binary measure where 0=no savings, 1=has savings) and total household savings amount. This measure evaluates household financial resilience and household capacity to accumulate and maintain financial reserves. Higher values indicate improved wealth accumulation and financial security.
Social safety net access at 2 months and 12 months | Baseline, 2 months, and 12 months
  Social safety net access is measured as a composite index assessing access to emergency financial support outside immediate household and close relatives. The index evaluates participants' ability to access 40 Philippine Pesos and 1,000 Philippine Pesos in emergency situations from extended social networks. The index is constructed using standardized methodology following Kling, Liebman, and Katz (2007), normalizing individual components against the control group before standardizing the aggregate measure. Higher scores indicate greater access to financial support networks.

CONTACTS AND LOCATIONS:
Overall Officials: Lincoln L Lau, PhD, Principal Investigator — University of Toronto; Melinda Kelly Mijares, MD, MPH, Principal Investigator — International Care Ministries; Tommy Lazaro III, MABE, PhD Candidate, Principal Investigator — Ateneo de Manila University

IPD SHARING:
Plan to Share IPD: Undecided
We are currently evaluating the feasibility of sharing individual participant data. Considerations include ethical approvals, participant consent, and the ability to sufficiently anonymize sensitive information. A final decision will be made in consultation with our ethics review board and institutional partners.

REFERENCES:
- [Background] Bryan G, Choi JJ, Karlan D. Randomizing religion: the impact of Protestant evangelism on economic outcomes. The Quarterly Journal of Economics. 2021 Feb;136(1):293-380.
- [Background] "Angrist, N., Kabay, S., Karlan, D., Lau, L., & Wong, K. (2025). Human Capital at Home: Evidence from a Randomized Evaluation in the Philippines (No. w33574). National Bureau of Economic Research.